CLINICAL TRIAL: NCT05469906
Title: Evaluation at 5 and 10 Years of Renal Transplant Patients Who Received a Graft Preserved in a Solution HEMO2life®
Brief Title: Evaluation at 5 and 10 Years of Renal Transplant Patients
Acronym: OXYOP 5 and 10
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OXYOP 5 and 10 (29BRC22.0144)
Record Dates: First submitted 2022-07-04; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Transplant; Complication, Failure
Keywords: renal transplantation; organ preservation; oxygen carrier

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interventional group: kidney graft preserved with M101
- control group: kidney graft preserved in standard condition (without M101)

SUMMARY:
5 and 10 years follow-up of the oxyop study.

DETAILED DESCRIPTION:
Oxyop (NCT02652520 PHRC) was a safety study evaluating the use of an oxygen carrier HEMO2life® as an additive in organ preservation solution in 60 transplanted kidneys. This was a national multicenter (6 centers) open-labeled safety study on HEMO2life® that included 58 recipients. The first patient was included on March 24th, 2016 and the study was completed on February 23th, 2018 (1 year of recruitment and 1 year of follow-up). Some efficacy secondary end points using a paired analysis was also analyzed (local kidney receiving HEMO2life® versus contralateral kidney transplanted elsewhere in France). Oxyop 5 and 10 years aims to analyse 5 and 10 years results.

ELIGIBILITY:
Inclusion Criteria:

* informed patients participating to the oxyop study
* Patient having completed the OXYOP M12 follow-up visit
* Patient agreeing to participate in the observational study

Exclusion Criteria:

* Opposition to the use his medical data
* patient deceased or with graft lost before M48

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 116 patients previously included in the oxyop study
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
eGFR | 10 years
  estimated GFR (CKDEPI)

SECONDARY OUTCOMES:
patient survival | 5 and 10 years
  patient survival at last follow-up
graft survival | 5 and 10 years
  graft survival at last follow-up
rejection rate | 5 and 10 years
  biopsy proven rejection
infection rate | 5 and 10 years
  all infection episodes
hospitalization | 5 and 10 years
  number of hospitalization, hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Le Meur, Principal Investigator — University hospital Brest France
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending five years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement